CLINICAL TRIAL: NCT06037980
Title: A Phase II/III Randomized Clinical Trial of CisPlatin plUs Gemcitabine and Nabpaclitaxel (GAP) as pReoperative Chemotherapy Versus Immediate Resection in patIents With resecTable BiliarY Tract Cancers (BTC) at High Risk for Recurrence: PURITY Study
Brief Title: CisPlatin plUs Gemcitabine and Nabpaclitaxel (GAP) as pReoperative Chemotherapy Versus Immediate Resection in patIents With resecTable BiliarY Tract Cancers (BTC) at High Risk for Recurrence
Acronym: PURITY
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PURITY
Record Dates: First submitted 2023-08-09; First posted 2023-09-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma
Keywords: Biliary Tract Cancers; Cholangiocarcinoma; Neoadjuvant Chemotherapy; Cisplatin Gemcitabine Nabpaclitaxel
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, multicenter, randomized phase II-III study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative chemotherapy (Experimental): Triplet combination of gemcitabine, cisplatin and nabpaclitaxel as neoadjuvant treatment followed by surgery and adjuvant chemotherapy
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: Cisplatin; Procedure: Curative Surgery; Drug: Capecitabine
- Upfront surgery (Active Comparator): Standard upfront surgery and adjuvant chemotherapy
  Interventions: Procedure: Curative Surgery; Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — ◦ Gemcitabine 800 mg/mq iv, day 1 and 8 of 21-day cycles, for 3 cycles
  Arms: Preoperative chemotherapy
Drug: Nab paclitaxel — ◦ Nab-paclitaxel 100 mg/mq, day 1 and 8 of 21-day cycles, for 3 cycles
  Other Names: Abraxane
  Arms: Preoperative chemotherapy
Drug: Cisplatin — ◦ Cisplatin 25 mg/mq iv, day 1 and 8 of 21-day cycles, for 3 cycles
  Arms: Preoperative chemotherapy
Procedure: Curative Surgery — Curative surgery on primary tumor
Drug: Capecitabine — 1250 mg/m2 given orally twice daily on days 1 to 14 of a 3 weekly cycle for a total of 8 cycles

SUMMARY:
PURITY is a multicentre, randomized adaptive phase II/III trial aimed at comparing the triplet combination of gemcitabine, cisplatin and nabpaclitaxel as neoadjuvant treatment (ARM A) versus standard upfront surgery (ARM B) in terms of 12-month PFS rate (phase II part) and PFS (phase III part) in patients with resectable BTC at high risk for recurrence.

DETAILED DESCRIPTION:
PURITY is a multicentre, randomized adaptive phase II/III trial aimed at comparing the triplet combination of gemcitabine, cisplatin and nabpaclitaxel as neoadjuvant treatment (ARM A) versus standard upfront surgery (ARM B) in terms of 12-month PFS rate (phase II part) and PFS (phase III part) in patients with resectable BTC at high risk for recurrence.

High risk for recurrence, for which patients will be eligible for study, is defined by the presence of at least one of the following risk features, as evaluated at baseline (pre-surgery):

1. For cholangiocarcinoma:

   * Suspected or definite locoregional lymph node involvement in the absence of jaundice (at least one of the following):

     * positive FNA cytology (obtained by EUS).
     * positive locoregional lymph nodes at PET-CT.
     * suspected positive locoregional lymph nodes at imaging (CT or MRI scan) according to local MTD discussion (eg. short axis > 1.5 cm, contrast enhancement uptake, round shape, restriction at DWI).
   * Macrovascular invasion at preoperative CT scan.
   * Expected R1 resection due to proximity to major intrahepatic vascular and biliary structures.
   * For iCCA, presence of satellitosis or multifocal disease or radiological suspicion of tumoral diaphragmatic adhesion.
   * For iCCA, size of the liver lesion >5 cm.
   * For eCCA, size of the primary lesion > 3cm.
   * Ca19.9 >100 U/mL.
2. For GBC:

   * Incidentally Detected Gallbladder Carcinoma (IGBC) After Simple Cholecystectomy with indication for radical second surgery (>pT2) or newly diagnosed GBC.

ELIGIBILITY:
Inclusion Criteria:

1. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures.
2. Female and male patients ≥18 years and <75 years.
3. Histologically or cytologically confirmed non metastatic resectable carcinoma of biliary tract (BTC), including gallbladder carcinoma (GBC), intrahepatic, periperihilar or distal Cholangiocarcinoma (CCA). Mixed tumor entities with hepatocellular carcinoma and ampullary cancers are excluded.
4. Availability of a tumoral sample
5. ECOG performance status of 0-1.
6. No prior tumor resection for BTC.
7. Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax and PET scan.
8. Technically resectable BTC as per local Multidisciplinary Team (MDT) assessment, including a core team with at least one medical oncologist, one surgeon, one radiologist, one endoscopist/gastroenterologist and one pathologist, all with expertise > 3 years on biliary tract cancer and hepatobiliary oncology.
9. High risk for recurrence defined as the presence of at least one of the following risk features, as evaluated at baseline (pre-surgery):

   1. For cholangiocarcinoma:

      * Suspected or definite locoregional lymph node involvement (at least one of the following):

        * positive FNA cytology (obtained by EUS).
        * positive locoregional lymph nodes at PET-CT.
        * suspected positive locoregional lymph nodes at imaging (CT or MRI scan) according to local MDT discussion (eg. short axis > 1.5 cm, contrast enhancement uptake, round shape, restriction at DWI).
      * Macrovascular invasion at preoperative CT scan.
      * Expected R1 resection due to proximity to major intrahepatic vascular and biliary structures.
      * For iCCA, presence of satellitosis or multifocal disease or radiological suspicion of tumoral diaphragmatic adhesion.
      * For iCCA, size of the liver lesion >5 cm.
      * For eCCA, size of the primary lesion > 3cm.
      * Ca19.9 >100 U/mL.
   2. For GBC:

      * Incidentally Detected Gallbladder Carcinoma (IGBC) after simple cholecystectomy with indication for radical second surgery (>pT2) or newly diagnosed GBC.
10. Estimated life expectancy > 3 months.
11. Adequate baseline hematologic function characterized by the following at screening:

    1. ANC ≥ 1.5 × 109/L
    2. platelets ≥ 100 × 109/L
    3. hemoglobin ≥ 9 g/dl. Note: prior transfusions for patients with low hemoglobin are allowed.
12. Adequate liver function characterized by the following at screening:

    1. Serum total bilirubin ≤ 1.5 × ULN and < 2 mg/dL. Note: Subjects with Serum total bilirubin ≥ 1.5 × ULN and conjugated bilirubin ≤ ULN or < 40% of total bilirubin are allowed.
    2. Serum transaminases (AST and/or ALT) < 3 x ULN.
13. Adequate renal function, i.e. serum creatinine ≤ 1.5 x institutional ULN and calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 50 mL/min
14. Adequate coagulation functions as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy).
15. No presence of complete dihydropyrimidine dehydrogenase (DPD) enzyme deficiency with DPYD gene testing mandatory at screening as per national guidelines
16. Females of childbearing potential must agree to remain abstinent (refrain from sexual intercourse) or use highly effective contraceptive methods, as defined in APPENDIX V of the full protocol, during the treatment period and for at least 7 months after the last administration of study treatments.
17. Males must agree to remain abstinent (refrain from sexual intercourse) or use highly effective contraceptive methods, as defined in APPENDIX V of the full protocol.
18. Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women <1 year after the onset of menopause.
19. A participant must agree not to donate eggs/sperm for future use for the purposes of assisted reproduction during the study and for a period of 7 months after receiving the last dose of study treatment. Female and male participants should consider preservation of eggs/sperm prior to study treatment as anti-cancer treatments may impair fertility.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any of the study drugs.
2. Any known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry except for curatively treated basal cell carcinoma of the skin, in situ carcinoma of the cervix, and prostate cancer.
3. Locally unresectable tumor according to local MDT (including radiological evidence suggesting inability to resect with curative intent whilst maintaining adequate vascular inflow and outflow, and sufficient future liver remnant).
4. Evidence of distant metastases at any site.
5. Tumors requiring multi-step surgical procedures such as two-stage hepatectomy or Associating Liver Partition and Portal vein Ligation for Staged hepatectomy (ALPPS) due to liver volumetry-based assessment of anticipated inadequate future liver remnant.
6. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic decompensation in the year before enrolment.
7. Know active uncontrolled hepatitis B or hepatitis C. Patients with a past or resolved HBV infection are eligible. Patients with chronic disease controlled by antiviral therapy or requiring prophylactic treatment are eligible.
8. Chronic or current active infectious disease requiring systemic antibiotics or antifungal treatment within 2 weeks prior to enrollment.
9. Known uncontrolled HIV infection. HIV-positive patients are eligible if their CD4+ cell count amounts to 300 cells per μL or more; HIV viral load must be undetectable per standard of care assay, and they must be compliant with antiretroviral treatment.
10. Pregnant or breast-feeding patient, or patient is planning to become pregnant within 7 months after the end of treatment.
11. Any other concurrent antineoplastic treatment including radiotherapy.
12. Previous or concurrent systemic (eg cytotoxic or targeted or other experimental drugs) therapy for BTC.
13. Prior surgery or locoregional therapy for BTC.
14. Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction in the last three months, significant arrhythmia).
15. Presence of psychiatric disorder precluding understanding of information of trial related topics and giving informed consent.
16. Any serious underlying medical conditions (judged by the investigator), that could impair the ability of the patient to participate in the trial.
17. Presence of complete dihydropyrimidine dehydrogenase (DPD) enzyme deficiency with DPYD gene testing mandatory at screening as per national guidelines.
18. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
12-month progression-free survival (PFS) rate | 12 months
  the proportion of patients alive and free from progression/post-resection recurrence by 12-months timepoint from randomization (to be considered as primary endpoint in the phase II part of the study and as secondary endpoint in the phase III part of the study).
median PFS | From date of randomization until the date of first documented progression (as assessed by radiological evaluation and clinical examination) or date of death from any cause, whichever came first, assessed up to 120 months
  i.e. the time from randomization to disease progression, post-resection recurrence or death from any cause (to be considered as secondary endpoint in the phase II part of the study and as primary endpoint in the phase III part of the study).

SECONDARY OUTCOMES:
Median event free survival | from date of randomization to disease progression that precludes definitive surgery, treatment discontinuation for any reason, post-resection recurrence, diagnosis of second cancer, or death from any cause, assessed up to 120 months
  i.e. the time from randomization to disease progression that precludes definitive surgery, treatment discontinuation for any reason, post-resection recurrence, a second primary cancer, or death from any cause.
Median relapse free survival | from date of surgery to date of disease recurrence or date of death, whichever came first, in patients who undergo surgery with curative intent, assessed up to 120 months.
  i.e. the time from surgery to disease recurrence or death in patients who undergo to surgery with curative intent.
Median Overall survival | from date of randomization to date of death (or last follow up for alive patients), assessed up to 120 months.
  i.e. the time from randomization to death or last follow-up for alive patients.
R0 resection rate | At surgery
  i.e. the percentage of patients, relative to the total of randomized patients, for whom a R0 resection is achieved.
R0+R1 resection rate | At surgery
  i.e. the percentage of patients, relative to the total of randomized patients, for whom the tumor was macroscopically removed and the intent of surgery is considered curative.
Quality of life EORTC QLQ-C30 scores | Quality of life questionnaires will be compiled during screening (28 days before randomisation) and at restaging before (week 8 to 10 after randomisation) and after surgery (week 6 to 16 after surgery)
  QoL will be estimated with EORTC QLQ-C30; mean score changes from baseline, proportion of patients with improved, stable, or deteriorated scores from baseline and time to deterioration in the EORTC QLQ-C30 scores will be compared between the two arms. Time to deterioration will be defined as the time from baseline to the first onset of a 10-point or greater decrease (for functional scales)/increase (for symptoms scale) from baseline, with confirmation under the right-censoring rule. All available observations will be used to calculate time to deterioration.
Quality of life BIL21 scores | Quality of life questionnaires will be compiled during screening (28 days before randomisation) and at restaging before (week 8 to 10 after randomisation) and after surgery (week 6 to 16 after surgery)
  QoL will be estimated with the module BIL21; mean score changes from baseline, proportion of patients with improved, stable, or deteriorated scores from baseline and time to deterioration in the BIL21 physical functioning, social functioning, and fatigue scores will be compared between the two arms. Time to deterioration was defined as the time from baseline to the first onset of a 10-point or greater decrease from baseline for functional scales or a 10-point or greater increase for symptom scales, with confirmation under the right-censoring rule. All available observations will be used to calculate time to deterioration.
Overall response rate | At radiological evaluation as performed at restaging before surgery (week 8 to 10 after randomisation)
  of neoadjuvant therapy as per investigator assessment and central review, i.e. the percentage of patients, relative to the total of enrolled subjects receiving neoadjuvant treatment, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria.
Resectability rate of primary tumor | Resectability rate will be assessed before surgery (after the 3 cycles of neoadjuvant chemotherapy for the experimental treatment arm)
  i.e. the retrospective evaluation of patients with unresectable disease, as assessed by the central review committee, in the two arms, and of the rate of conversion to resectability in the neoadjuvant arm.
Toxicity rates | Through study completion, an average of 1 year for each patient
  .e. the percentage of patients, relative to the total of subjects randomized to neoadjuvant treatment, experiencing a specific adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0).
Perioperative morbidity and mortality | At surgery
  i.e. the percentage of patients, relative to the total of enrolled subjects undergoing surgery, with any serious perioperative morbidity or mortality according to Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Niger, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Monica Niger, MD, Principal Investigator — 02 2390 2919
Locations (19):
- Italy (19):
  - Ospedali Riuniti di Ancona, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Oncologia Medica Policlinico Sant'Orsola - Malpighi, Bologna
  - ASST Spedali Civili, Brescia
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - IRST Dino Amadori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Humanitas Cancer Center, Milan
  - Ospedale Niguarda Cancer Center, Milan
  - Ospedale San Raffaele, Milan
  - Università di Modena, Modena
  - Ospedale S. Gerardo, Monza
  - IOV, Padua
  - Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Pisa, Pisa
  - IRST (Cesena-Forlì-Meldola), Ravenna
  - Policlinico Gemelli, Rome
  - Azienda Ospedaliera Ordine Mauriziano, Turin
  - AOUI Verona - Policlinico "G.B. Rossi", Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yadav S, Xie H, Bin-Riaz I, Sharma P, Durani U, Goyal G, Borah B, Borad MJ, Smoot RL, Roberts LR, Go RS, McWilliams RR, Mahipal A. Neoadjuvant vs. adjuvant chemotherapy for cholangiocarcinoma: A propensity score matched analysis. Eur J Surg Oncol. 2019 Aug;45(8):1432-1438. doi: 10.1016/j.ejso.2019.03.023. Epub 2019 Mar 21. PMID 30914290
- [Result] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Result] Maithel SK, Keilson JM, Cao HST, Rupji M, Mahipal A, Lin BS, Javle MM, Cleary SP, Akce M, Switchenko JM, Rocha FG. NEO-GAP: A Single-Arm, Phase II Feasibility Trial of Neoadjuvant Gemcitabine, Cisplatin, and Nab-Paclitaxel for Resectable, High-Risk Intrahepatic Cholangiocarcinoma. Ann Surg Oncol. 2023 Oct;30(11):6558-6566. doi: 10.1245/s10434-023-13809-5. Epub 2023 Jun 27. PMID 37368098
- [Derived] Niger M, Nichetti F, Fornaro L, Pircher C, Morano F, Palermo F, Rimassa L, Pressiani T, Berardi R, Gardini AC, Sperti E, Salvatore L, Melisi D, Bergamo F, Siena S, Mosconi S, Longarini R, Arcangeli G, Corallo S, Delliponti L, Tamberi S, Fea E, Brandi G, Rapposelli IG, Salati M, Baili P, Miceli R, Ljevar S, Cavallo I, Sottotetti E, Martinetti A, Busset MDD, Sposito C, Di Bartolomeo M, Pietrantonio F, de Braud F, Mazzaferro V. A phase II/III randomized clinical trial of CisPlatin plUs Gemcitabine and Nabpaclitaxel (GAP) as pReoperative chemotherapy versus immediate resection in patIents with resecTable BiliarY Tract Cancers (BTC) at high risk for recurrence: PURITY study. BMC Cancer. 2024 Apr 8;24(1):436. doi: 10.1186/s12885-024-12225-6. PMID 38589856